CLINICAL TRIAL: NCT01378468
Title: The Berlin 'Cream&Sugar' Study: the Prognostic Impact of an Oral Triglyceride Tolerance Test in Patients After Acute Ischemic Stroke
Brief Title: Prognostic Impact of an Oral Triglyceride Tolerance Test in Patients After Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Martin Ebinger, PD Dr. med. Dr. phil., Charite University, Berlin, Germany
Other Study IDs: The Berlin 'Cream&Sugar' Study; 2009-010356-97 (EudraCT Number)
Record Dates: First submitted 2011-06-21; First posted 2011-06-22 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: First Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with first ischemic stroke
  Interventions: Other: oral triglyceride tolerance test (not a therapeutic "intervention" as such but a new diagnostic test)

INTERVENTIONS:
Other: oral triglyceride tolerance test (not a therapeutic "intervention" as such but a new diagnostic test) — see Ebinger et al., IJS, 2010
  Other Names: cream

SUMMARY:
Non-fasting triglyceride levels are thought to play a role in stroke. The investigators hypothesise that the results of a standardised oral triglyceride tolerance test in the subacute setting (3-7 days) after the first ischaemic stroke are associated with the risk of recurrent stroke within 12 months after the index event.

DETAILED DESCRIPTION:
Since high postprandial triglycerides levels may be a risk factor for stroke, we use a combined oral triglyceride and glucose tolerance test in patients who had a first ischemic stroke. Follow-up after one year primarily assesses wether or not a recurrent stroke has occured. The glucose tolerance test is meant to identify patients with metabolic syndrome (and diabetes), since this condition is per se associated with increased levels of triglycerides. Potentially, the post-challenge triglyceride levels only play a role in patients without diabetes or metabolic syndrome. For further details see Ebinger et al. 'The Berlin 'Cream&Sugar' Study: the prognostic impact of an oral triglyceride tolerance test in patients after acute ischaemic stroke', IJS; 2010,5, 47-51.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* First ischemic stroke
* Incidence within less than 7 days
* Informed consent obtained

Exclusion Criteria:

* Aphasia (if hampering informed consent)
* Swallowing disorder
* Pregnancy
* Renal or hepatic failure
* Pancreatitis
* Cholecystolithiasis
* Malabsorption
* Lactose intolerance
* Psychosis
* Drug and/or alcohol addiction
* Expected life expectancyr12 months
* Inability to sign informed consent
* Acute coronary syndrome
* Severe heart valve disorder
* Heart failure (NYHA III-IV)
* Severe infectious/rheumatic disease
* Sever metabolic disease
* No oral glucose tolerance test in case of known diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study population consists of adults with first ischemic stroke within the last three to seven days (at time of testing).
Sampling Method: Non-Probability Sample
Enrollment: 573 (Actual)
Dates: Start 2009-01; Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Recurrent Stroke | outcome measure is assessed one year after first ischemic stroke.
  The primary end-point of the study is a recurrent fatal or nonfatal stroke within the first 12 months after the event.

SECONDARY OUTCOMES:
MI | one year after first ischemic stroke
  Myocardial infarction
death | one year after first ischemic stroke
  cardiovascular death (death due to any cardiovascular or cerebrovascular event)
TIA | one year after first ischemic stroke
  transient ischemic attack

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ebinger, Principal Investigator — CSB; Matthias Endres, Principal Investigator — CSB
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Ebinger M, Heuschmann PU, Jungehuelsing GJ, Werner C, Laufs U, Endres M. The Berlin 'Cream&Sugar' Study: the prognostic impact of an oral triglyceride tolerance test in patients after acute ischaemic stroke. Int J Stroke. 2010 Apr;5(2):126-30. doi: 10.1111/j.1747-4949.2010.00399.x. PMID 20446947
- [Derived] Lange KS, Nave AH, Liman TG, Grittner U, Endres M, Ebinger M. Lipoprotein(a) Levels and Recurrent Vascular Events After First Ischemic Stroke. Stroke. 2017 Jan;48(1):36-42. doi: 10.1161/STROKEAHA.116.014436. Epub 2016 Nov 17. PMID 27856951
- [Derived] Batluk J, Leonards CO, Grittner U, Lange KS, Schreiber SJ, Endres M, Ebinger M. Triglycerides and carotid intima-media thickness in ischemic stroke patients. Atherosclerosis. 2015 Nov;243(1):186-91. doi: 10.1016/j.atherosclerosis.2015.09.003. Epub 2015 Sep 9. PMID 26398290
- [Derived] Leonards CO, Ipsen N, Malzahn U, Fiebach JB, Endres M, Ebinger M. White matter lesion severity in mild acute ischemic stroke patients and functional outcome after 1 year. Stroke. 2012 Nov;43(11):3046-51. doi: 10.1161/STROKEAHA.111.646554. Epub 2012 Aug 30. PMID 22935398